CLINICAL TRIAL: NCT05039372
Title: The Effect Of Nurse Counselıng Applıed Accordıng To Planned Behavıor Theory On Paın, Fatıgue And Functıonal Status In Patıents Wıth Rheumatoid Arthritis
Brief Title: Rheumatoid Arthritis, Planned Behavıor Theory And Nurse Counselıng
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Keriman Aytekin Kanadli, Principal Investigator, Hasan Kalyoncu University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: interventional
Record Dates: First submitted 2021-09-02; First posted 2021-09-09 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Planned Behavior Theory
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: experimental randomized controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- training and consultancy (Experimental): "Patient Description Form, Bristol Rheumatoid Arthritis Fatigue Multidimensional Questionnaire, McGill Pain Scale Short Form, Stanford Health Assessment Questionnaire" will be administered to the patients in this group at the first interview. Individual training will be given to the patient in line with the training guide prepared for the rheumatoid arthritis patient, and the guide will be shared after the training. In line with the theory of planned behavior in patients with rheumatoid arthritis, counseling service will be provided by the researcher to the extent of the training plan prepared for symptom management. At the end of the 3rd month, the patients will be interviewed face to face and the "Bristol Rheumatoid Arthritis Fatigue Multidimensional Questionnaire, McGill Pain Scale Short Form, Stanford Health Assessment Questionnaire" will be administered again.
  Interventions: Behavioral: TRAINING AND CONSULTANCY
- control (No Intervention): After obtaining written consent from the patients who agreed to participate in the study, the patients included in the control group were asked to continue their rheumatologist follow-up and their normal lives (hospital routine, daily life). Patients in this group will fill out the "Patient Description Form, Bristol Rheumatoid Arthritis Fatigue Multidimensional Questionnaire, McGill Pain Scale Short Form, Stanford Health Evaluation Questionnaire" at the first interview. After 3 months, data collection tools other than the "Patient Identification Form" will be applied to the patients and the training guide to be prepared for rheumatoid arthritis patients will be given.

INTERVENTIONS:
Behavioral: TRAINING AND CONSULTANCY — TRAINING AND CONSULTANCY
  Arms: training and consultancy

SUMMARY:
Ensuring disease management begins with comprehensive education and drug therapy. Symptoms such as deformities, pain and fatigue, which are most common in rheumatoid arthritis patients, seriously affect the daily activities of the patients. In order to improve the quality of life of the patient, it is essential that he receives planned education about his disease and constant follow up it like this helps him manage his disease by providing behavioral changes. There are similar studies on chronic diseases in the literature, and it has been seen to make a positive contribution. Studies have shown that patient education includes only information, counseling or behavioral therapies, and does not necessarily turn into behavior change on its own. Which was developed on the basis of education and human behavior theories, According to The Theory of Planned Behavior it is thought that patients can cope with their illnes, manage their illnesses and show behavioral changes by adapting to the illness with the help of nursing counseling. The importance of patient follow-up has once again come to the fore when it comes to the problems that those with chronic diseases may experience during the pandemic process and the difficulties in finding solutions. Recently, training and follow-up are carried out with remote access in the management of many chronic diseases. Especially in chronic diseases such as rheumatoid arthritis, which affects all systems, the counseling service to be provided to the extent that behavior change can be achieved has become more important. In this direction, it is thought that it will be beneficial in the long term for patients to gain behavioral changes by telephone monitoring after education.

DETAILED DESCRIPTION:
Examining the studies in the literature, the effect size between the experimental group and the control group was calculated and it was estimated to be around 0.70. In the experimental and control groups, a total of 68 individuals, including at least 34 individuals in both groups, should be included in the study in order to determine the difference between the groups in the power analysis calculated with 80% power and 0.05 significance. Considering that there would be individuals who could not continue to work or could not be reached afterwards, the number of required to be reached individuals was calculated as 74 individuals. In this study, the sample size was calculated with the GPower program version 3.1.

Type and Time of Research

This research is planned to be conducted as a randomized controlled experimental study.

Application of Research

In the research, the applications to be made to the control and experimental groups are explained separately:

*Control Group Intervention: After obtaining written consent from the patients who agreed to participate in the study, the patients included in the control group were asked to continue their rheumatologist follow-up and their normal lives (hospital routine, daily life). Patients in this group will fill out the "Patient Description Form, Bristol Rheumatoid Arthritis Fatigue Multidimensional Questionnaire, McGill Pain Scale Short Form, Stanford Health Evaluation Questionnaire" at the first interview. After 3 months, data collection tools other than the "Patient Identification Form" will be applied to the patients and the training guide to be prepared for Rheumatoid Arthritis patients will be given.

Experimental Group Initiative: After obtaining written consent from the patients who agreed to participate in the study, they will be asked to continue with their rheumatologist follow-up and their normal lives (hospital routine, daily life).

"Patient Description Form, Bristol Rheumatoid Arthritis Fatigue Multidimensional Questionnaire, McGill Pain Scale Short Form, Stanford Health Assessment Questionnaire" will be administered to the patients in this group at the first interview. Individual training will be given to the patient in line with the training guide prepared for the rheumatoid arthritis patient, and the guide will be shared after the training. Mutual contact information will be shared with the patient and it will be stated that he can call during the counseling period (3 months).In line with the theory of planned behavior in patients with Rheumatoid Arthritis counseling service will be provided by the researcher to the extent of the training plan prepared for symptom management. At the end of the 3rd month, the patients will be interviewed face to face and the "Bristol Rheumatoid Arthritis Fatigue Multidimensional Questionnaire, McGill Pain Scale Short Form, Stanford Health Assessment Questionnaire" will be administered again.

ELIGIBILITY:
Criteria:

Inclusion Criteria for Research

* Between 18 and 64 years old
* Diagnosed with Rheumatoid Arthritis at least 6 months ago,
* Can communicate in Turkish and does not have a cognitive problem that prevents communication,
* No neurological or psychiatric disease without malignancy,
* Without heart failure (stages III and IV according to NYHA)
* Not pregnant,
* Able to use a telephone,
* Patients who volunteer to participate in the study will be included in the study.

Exclusion Criteria

* Under 18 years old,
* Newly diagnosed, treated for less than 6 months,
* Having a malignant type of disease,
* Patients who do not volunteer to participate in the study will not be included.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2022-01-30 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of Patient-Reported Fatigue | 0-3 months
  Bristol Rheumatoid Arthritis Fatigue Multidimensional Questionnaire (BRAF-MDQ): It was developed to evaluate the effect of fatigue in different dimensions in patients with rheumatoid arthritis. There are 20 questions in total. Total BRAF-MDQ scores range from 0 to 70. Higher scores indicate higher fatigue.
Evaluation of Patient-Reported Pain | 0-3 months
  McGill Pain Scale Short Form (MAS-SF): The scale provides information about the sensory characteristics, severity and effect of pain. The main component of the scale consists of 15 descriptive adjectives for sensation of pain and is self-rated by the patient according to the level of intensity on a scoring scale (0 = none, 1 = mild, 2 = moderate, 3 = severe).
Assessment of Patient-Reported Functional Status | 0-3 months
  Stanford Health Assessment Scale (HAQ): The Health Assessment Scale is a functional measurement method that is frequently used to evaluate the functional status of rheumatology patients in their daily lives. The scale consists of 20 items in the form of 8 sections. A high score on the scale indicates functional disability.

CONTACTS AND LOCATIONS:
Overall Officials: Nermin Olgun, professor, Study Director — Hasan Kalyoncu University Faculty of Nursing
Locations (1):
- Hasan Kalyoncu Uninersity, Gaziantep, Turkey (Türkiye)